CLINICAL TRIAL: NCT03819881
Title: A Phase 1b, Multi-centered, Randomized, Double-blind, Placebo-controlled, Parallel Group, Three Sequential Part Study of STMC-103H in Multi-Sensitized Allergic Subjects Who Are Otherwise Healthy
Brief Title: A Phase 1b Study of STMC-103H in Multi-Sensitized Allergic Subjects Who Are Otherwise Healthy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Siolta Therapeutics, Inc. (Industry)
Collaborators: Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STMC-103H-101
Record Dates: First submitted 2019-01-10; First posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Atopic Immunoglobulin E-Mediated Allergic Disorder

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two arms in three sequential age-descending cohorts:
  Part 1: 18-40 years of age Part 2: 12-17 years of age Part 3: 2-11 years of age
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- STMC-103H (Experimental): Oral administration of STMC-103H twice daily, randomized 3:1 (STMC-103H:Placebo) in three age-descending groups:
  Part 1: 20 subjects 18-40 years of age Part 2: 20 subjects, 12-17 years of age Part 3: 20 subjects, 2-11 years of age
  Interventions: Biological: STMC-103H
- Placebo (Placebo Comparator): Oral administration of placebo twice daily, randomized 3:1 (STMC-103H:Placebo) in three age-descending groups:
  Part 1: 20 subjects 18-40 years of age Part 2: 20 subjects, 12-17 years of age Part 3: 20 subjects, 2-11 years of age
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: STMC-103H — Live bacterial product
  Arms: STMC-103H
Biological: Placebo — Inactive placebo substance
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of STMC-103H compared to placebo in allergic subjects who are otherwise healthy.

DETAILED DESCRIPTION:
This is a first-in-human trial of this live biotherapeutic product. The primary objective is to assess safety and tolerability in allergic subjects who are otherwise healthy, with twice daily dosing in descending age groups.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary informed consent from subject or legally acceptable representative and/or child assent from the subject (as applicable).
* For part 1, subjects of 18 years to 40 years of age at the timing of the signature on the informed consent.
* For part 2, subjects of 12 years to 17 years of age at the timing of the signature on the informed consent.
* For part 3, subjects of 2 years to 11 years of age at the timing of the signature on the informed consent.
* Good health and free of significant diseases or clinically significant abnormal findings on physical exam and laboratory evaluations.
* No history or presence of gastrointestinal, hepatic, or renal disease/disorder.
* History of allergic disease confirmed by 2 or more episodes in past 5 years.
* Positive skin prick test to two or more common allergens.
* Subjects who are of childbearing potential must agree to remain abstinent from heterosexual activity or agree to use (or have their partner use) acceptable contraception to prevent pregnancy within projected duration of the trial.

Exclusion Criteria:

* Presence or history of any significant acute or chronic medical illness, except for allergic disease.
* BMI > 32 kg/m2 at the time of signing consent.
* Current or persistent moderate to sever asthma that requires use of control medication (Step 3 or above, according to Asthma Step Program).
* Presence of rhinitis secondary to causes other than allergy.
* History of anaphylaxis.
* Any known allergies to two or more of the following three antibiotics: Augmentin, tetracycline, or bacitracin.
* Inability to be venipunctured and/or tolerate venous access (Parts 1 and 2 only).
* Consistent consumption of probiotics ≥ 2 days / week over multiple weeks within the 3 months prior to the study Baseline Visit.
* Regular use of any of the following medications:

  * Intranasal or systemic corticosteroids (in 1 month prior to screening or during study)
  * Leukotriene modifiers (in 1 month prior to screening or during study)
  * Intranasal cromolyn (in 2 weeks prior to screening or during study)
  * Intranasal or systemic decongestants (in 3 days prior to screening or during study)
  * Cetirizine, fexofenadine, loratadine, desloratadine, hydroxyzine (in 10 days prior to screening or during study)
  * Intranasal antihistamines (in 3 days prior to screening or during study)
  * Other systemic antihistamines (in 3 days prior to screening or during study)
* Allergies to excipients in the Investigational Product formulation.
* Allergy to soy in any form.
* Presently consuming alcohol more than 2 glasses per day or has history of alcohol dependence or alcohol abuse during the past one year prior to screening.
* Presently a smoker or ex-smoker with history of smoking (subject must abstain from smoking throughout the study).
* History or presence of significant recreational or illicit drug abuse in past 1 year.
* Participation in another clinical study within 30 days prior to screening.
* Use of any probiotic or prebiotic in the past 3 months prior to screening.

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients with treatment-related adverse events (AEs) assessed as mild, moderate and severe, from baseline to day 29. | From baseline to day 57
  All adverse events (AEs) recorded during the study through the date of randomization up to 28 days after the last dose of study drug will analyzed.
  Treatment-emergent AEs (TEAEs), defined as any AE that starts or increases in severity after the first dose of STMC-103H or placebo, will be summarized. The total number of reported AEs will also be summarized.
Incidence of abnormal laboratory test results from baseline to day 29 | From baseline to day 29
  The change in laboratory results from baseline to day 29 in multi-sensitized (to two or more allergens) subjects who are otherwise healthy and who have completed BID dosing of STMC-103H or placebo for 28 days
Change in blood pressure from baseline to day 57 | From baseline to day 57
  Observed values of blood pressure obtained at screening and study Days 1, 8, 15, 22, 29, 43, and 57) and corresponding changes from baseline (Day 1) will be listed and summarized by descriptive statistics by study part and visit.
Change in respiration rate from baseline to day 57 | From baseline to day 57
  Observed values of respiration rate obtained at screening and study Days 1, 8, 15, 22, 29, 43, and 57) and corresponding changes from baseline (Day 1) will be listed and summarized by descriptive statistics by study part and visit.
Change in heart rate from baseline to day 57 | From baseline to day 57
  Observed values of heart rate obtained at screening and study Days 1, 8, 15, 22, 29, 43, and 57) and corresponding changes from baseline (Day 1) will be listed and summarized by descriptive statistics by study part and visit.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Neutel, MD, Principal Investigator — Orange County Research Center
Locations (2):
- United States (2):
  - Bensch Clinical Research LLC, Stockton, California
  - Orange County Research Center, Tustin, California

IPD SHARING:
Plan to Share IPD: No